CLINICAL TRIAL: NCT01657110
Title: Uncontrolled, Open-label, Phase II Pilot Study to Evaluate the Efficacy, Tolerability and Acceptability of 200mg/g Tea Tree Oil Gel Applied Topically Twice Daily for the Treatment of Mild to Moderate Facial Acne
Brief Title: Pilot Study to Evaluate Tea Tree Oil Gel for Facial Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: Royal Perth Hospital (Other); Hollywood Private Hospital (Unknown)
Responsible Party: Principal Investigator, Katherine Hammer, Research Assistant Professor, The University of Western Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRJ-006245
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Acne
Keywords: acne; inflamed lesions; non-inflamed lesions; complementary medicine; essential oil
MeSH Terms: conditions — Acne Vulgaris | interventions — Tea Tree Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tea tree oil (Other): Pea-sized amount of tea tree oil medicated gel (containing 200mg/g tea tree oil) applied to the face twice daily for 12 weeks.
  Interventions: Other: Tea tree oil

INTERVENTIONS:
Other: Tea tree oil — Pea-sized amount of tea tree oil medicated gel (containing 200mg/g tea tree oil) applied to the face twice daily for 12 weeks.
  Other Names: melaleuca oil; Thursday Plantation

SUMMARY:
Mild to moderate facial acne is an extremely common disease of teenagers and young adults. This pilot study will investigate whether treatment with a gel containing tea tree oil reduces numbers of acne lesions and improves acne in twenty otherwise healthy consenting participants. The hypothesis is that treatment with tea tree oil gel will result in a significant improvement in acne after 12 weeks of treatment.

DETAILED DESCRIPTION:
Tea tree oil is the essential oil obtained from the Australian plant Melaleuca alternifolia. The oil has been used in Australia for many decades as a topically applied antiseptic and has been used to treat bites, stings, cuts and grazes. Many studies have shown that tea tree oil has both antimicrobial and anti-inflammatory activity in the laboratory. In addition, clinical trials have demonstrated that the oil can help in treating conditions such as dandruff, tinea, colonisation with methicillin resistant Staphylococcus aureus (MRSA) in the nose and acne. Together, these laboratory and clinical studies indicate that tea tree oil can potentially be used to treat relatively minor skin infections or diseases.

This pilot study aims to investigate whether a commercially available gel containing tea tree oil is effective for treating mild to moderate facial acne. A minimum of 18 participants that meet the inclusion and exclusion criteria will be enrolled in the study. Participants will be instructed to apply the tea tree oil gel each morning and night for 12 weeks and their acne will be assessed after 4, 8 and 12 weeks of treatment. Acne severity will be measured by (1) counting the numbers of lesions (pimples) on the face and (2) assigning an overall acne severity score. The lesion counts and severity scores at 4, 8 and 12 weeks will be compared to the baseline count to evaluate whether the acne is improving.

Potential benefits to participants, and of the study, are that their acne may improve as a result of treatment and that the results of the study may provide evidence that a commercially available product is effective for treating acne. There are many over-the-counter topically applied products available for treating acne. Two of the most common active ingredients are benzoyl peroxide and salicylic acid. Benzoyl peroxide is an antibacterial agent that works by killing the P. acnes bacterium on the skin. Although it is relatively effective for treating acne, it can also be quite irritating, especially when patients first start to use it. Salicylic acid acts by helping to unblock pores and remove excess dead skin thus helping pimples to heal more quickly. However, it is generally not as effective as benzoyl peroxide. One previous study has shown that a gel containing 5% tea tree oil performed similarly to benzoyl peroxide for reducing pimples, suggesting that it warrants further study.

Since a small percentage of people (approximately 1.4%) are allergic to tea tree oil all participants will be monitored for any reactions to the study product. Tea tree oil allergy typically manifests as redness and swelling and the site of application. This is one of the possible risks to participants, however, given the small numbers of study participants the likelihood of one or more participants having a reaction to the oil is low. Another possible risk is that participants may not benefit from the treatment and that their acne may not improve.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 - 45 years
2. Mild to moderate facial acne with 10 - 100 lesions
3. Investigator Global Assessment score of at least 2
4. Able to comply with the requirements of the protocol and attend the outpatients clinic at 2, 4, 8 and 12 weeks
5. Able to provide written informed consent

Exclusion Criteria:

1. More than 2 acne nodules
2. Allergy to tea tree oil or any component of the study drug
3. Current skin disease (other than acne)
4. Facial hair that may obscure acne lesions
5. Use of topical or systemic steroids within the last 2 or 4 weeks, respectively
6. Use of topical or systemic antibiotics within the last 2 or 4 weeks, respectively
7. Use of topical acne treatments (eg. benzoyl peroxide, salicylates, retinoids) within the last 2 weeks
8. Use of systemic retinoids within the past 6 months
9. Procedures on the face such as peels, laser therapy or microdermabrasion within the past 4 weeks
10. Women who are pregnant or breastfeeding
11. Women of childbearing potential not using a reliable contraceptive method. Participants taking oral contraceptives must have been taking their current contraceptive for the previous 3 months and must agree to continue with it until study completion.
12. Participation in another clinical trial during the last 12 weeks
13. Concurrent diseases which exclude the administration of therapy as outlined by the study protocol
14. Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study and/or likely to cause death within the study duration
15. Chronic lung disease with hypoxemia
16. Myocardial infarction during the last 6 months
17. Non-compensated heart failure
18. Severe non-compensated hypertension
19. Severe non-compensated diabetes mellitus
20. Severe psychiatric disease
21. Known HIV or active chronic hepatitis B or C infection
22. Subjects who, in the opinion of the investigator, are not likely to complete the study for what ever reason.
23. Subjects who, in the opinion of the investigator, abuse alcohol or drugs

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Lesion numbers | 12 weeks
  Numbers of inflamed and non-inflamed facial lesions will be counted.
Investigator Global Assessment | 12 weeks
  A 5-point severity scale (0-4) will be used to give an overall acne grade.
  0: Clear skin with no lesions
  1. Almost clear; rare lesions
  2. Mild severity; some non-inflammatory lesions with no more than a few inflammatory lesions
  3. Moderate severity; up to many non-inflammatory lesions and may have some inflammatory lesions
  4. Severe; up to many noninflammatory and inflammatory lesions but no more than a few nodular lesions

SECONDARY OUTCOMES:
Decreased non-inflammatory lesion count | 12 weeks
  Decrease in numbers of non-inflammatory lesions from baseline
Decreased inflammatory lesion count | 12 weeks
  Decrease in inflammatory lesion count from baseline
Decrease in perceived facial oiliness | 12 weeks
  Decrease in perceived facial oiliness from baseline

OTHER OUTCOMES:
Mean tolerability score | 12 weeks
  Mean tolerability will be determined as the average of the following;
  1. Erythema
  2. Scaling
  3. Peeling
  4. Burning
  5. Induration
  6. Dryness
  These six parameters will be measured using a 5-point scale (0: None, 1: Minimal, 2: Mild, 3: Moderate, 4: Severe). Mean tolerability will be the average of these scores.
The frequency of adverse events | 12 weeks
  Any local or systemic adverse events will be recorded including the type of reaction and severity (on a 5-point severity scale where 0 = none and 4 = severe).

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Kumarasinghe, Principal Investigator — Royal Perth Hospital
Locations (2):
- Australia (2):
  - Royal Perth Hospital, Perth, Western Australia
  - Hollywood Private Hospital, Perth

REFERENCES:
- [Background] Carson CF, Hammer KA, Riley TV. Melaleuca alternifolia (Tea Tree) oil: a review of antimicrobial and other medicinal properties. Clin Microbiol Rev. 2006 Jan;19(1):50-62. doi: 10.1128/CMR.19.1.50-62.2006. PMID 16418522